CLINICAL TRIAL: NCT03711435
Title: Study on TCM Syndrome Classification of Idiopathic Pulmonary Fibrosis Based on Metabolomics
Brief Title: Traditional Chinese Medicine(TCM) Syndrome Classification of Idiopathic Pulmonary Fibrosis(IPF) and Metabolomics
Status: Completed | Type: Observational
Sponsor: Xuzhou Traditional Chinese Medicine Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XZTCM2018LSY-013
Record Dates: First submitted 2018-10-07; First posted 2018-10-18 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Metabolomics; Chinese medicine
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood

GROUPS / COHORTS (2):
- Training set: The training set is composed of 30 IPF patients and 15 controls. The group is designed to identify differential metabolites between IPF and control groups.
- Validation set: The validation set is composed of 15 IPF patients and 15 controls. The group is designed to validate differential metabolites identified in the previous groups.

SUMMARY:
The pathogenesis of idiopathic pulmonary interstitial fibrosis is complex, and there is no specific biomarkers, the treatment effect is not such useful. Currently, it is discovered that Chinese medicine treatment may be effective. The investigators select patients with idiopathic pulmonary interstitial fibrosis and healthy controls, use metabolomics to study the biological characteristics of idiopathic pulmonary interstitial fibrosis, screen biomarkers of IPF, and label different TCM syndromes of IPF, explore the biological nature of IPF TCM syndromes, find the biological changes that occur during the development and progression of IPF and explore the metabolite marker clusters of IPF. Furthermore, the results of this study may find its diagnostic significance for IPF and Looking for potential targets for future treatment of IPF.

ELIGIBILITY:
Inclusion Criteria:

* Case group inclusion criteria

  1. According to the diagnostic criteria published in 2015, the New Guidelines for the Diagnosis and Treatment of Idiopathic Pulmonary Fibrosis, jointly developed by the American Thoracic Society, the European Respiratory Society, the Japanese Respiratory Society, and the Latin American Thoracic Society;
  2. aged 50 to 85 years old;

Control group inclusion criteria:

Health people match on the age (±3 years old) and gender with case group with 1:1 rate at the same time.

Exclusion Criteria:

* Case group exclusion criteria:

  1. Those with severe heart, liver, kidney and other organ dysfunction or suffering from blood diseases;
  2. with malignant tumors;
  3. Severely infected people;
  4. Pregnant and lactating women;
  5. mental illness, serious obstacles and those who are unwilling to cooperate;

Control group exclusion criteria:

1. Those with severe heart, liver, kidney and other organ dysfunction or blood disease;
2. With malignant tumors;
3. Chest X-ray or chest low-dose CT suggesting intra-pulmonary interstitial fibrosis;
4. With chronic pulmonary diseases such as pulmonary interstitial disease, chronic obstructive pulmonary disease, and bronchial asthma;
5. With connective tissue disease and those with a history of exposure to occupational diseases;
6. Mental illness, serious obstacles and unwilling to cooperate.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IPF patients in XUZHOU
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
biomarkers detected in metabolites | 1 year
  Metabolomics of serum based on mass spectrometry.It is non-targeted metabolomics.The study is to find the target metabolite to distinguish IPF.

SECONDARY OUTCOMES:
High-resolution chest CT total score (CT-Tot) | 1 year
  High-resolution chest CT total score (CT-Tot), which includes the grid shadow and the honeycomb lung. The score range is 0-5, and the larger the score, the more serious the disease.
Six Minute Walk Test(6MWT) | 1 year
  The six-minute walk test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface.It is a simple objective indicator for evaluating cardiopulmonary function
Pulmonary function Pulmonary function | 1 year
  Pulmonary function including forced vital capacity(FVC),forced expiratory volume at one second(FEV1),diffusion capacity of lung for carbon monoxide(DLCO)
St. George's Respiratory Questionnaire | 1 year
  St. George's Respiratory Questionnaire is measuring impaired health and perceived well-being ('quality of life') in airways disease. the score is 0 to 100，the higher the score is，the worse life quality the patients has.

CONTACTS AND LOCATIONS:
Overall Officials: YING MS ZHAO, PHD, Principal Investigator — Xuzhou Traditional Chinese Medicine Hospital
Locations (1):
- Xuzhou Traditional Chinese Medicine Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Other researchers may contact us with email